CLINICAL TRIAL: NCT00648154
Title: Single-Dose Fed Bioequivalence Study of Letrozole Tablets (2.5 mg; Mylan) and Femara® Tablets (2.5 mg; Novartis) in Healthy Postmenopausal Female Volunteers
Brief Title: Food Study of Letrozole Tablets 2.5 mg and Femara® Tablets 2.5 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Wayne Talton, Mylan Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LETR-05123
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
MeSH Terms: interventions — Letrozole

ARMS (2):
- 1 (Experimental): Letrozole Tablets 2.5 mg
  Interventions: Drug: Letrozole Tablets 2.5 mg
- 2 (Active Comparator): Femara® Tablets 2.5 mg
  Interventions: Drug: Femara® Tablets 2.5 mg

INTERVENTIONS:
Drug: Letrozole Tablets 2.5 mg — 2.5mg, single dose fed
  Arms: 1
Drug: Femara® Tablets 2.5 mg — 2.5mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's letrozole 2.5 mg tablets to Novartis' Femara® 2.5 mg tablets following a single, oral 2.5 mg (1 x 2.5 mg) dose administered under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 40 years or older.
2. Sex: Females only.
3. Weight: At least 52 kg (115 lbs) and within 30% of Ideal Body Weight (IBW), as referenced by the Table of ""Desirable Weights of Adults"" from Metropolitan Life Insurance Company, 1999 (See Part II: ADMINISTRATIVE ASPECTS OF HUMAN BIOAVAILABILITY PROTOCOLS).
4. Absence of menses for one year for postmenopausal subjects, or at least 6 weeks for oophorectomized subjects. (For oophorectomized subjects, an operative report documenting bilateral oophorectomy and surgical pathology report documenting the absence of malignant disease.)
5. Baseline FSH and 17β-estradiol serum levels consistent with postmenopausal status confirmed within 72 hours of initiation of study medication (FSH greater than or equal to 40 mIU/mL; 17β-estradiol less than or equal to 31 pg/mL).
6. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, 12-lead ECG, Hepatitis B, Hepatitis C and HIV tests, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiates, phencyclidine, and methadone) performed within 21 days of the initial dose of study medication.
7. The physical examination shall include pelvic and breast exams.

   1. Pelvic findings should be consistent with hypoestrogenemia.
   2. A mammogram will be required if not performed within the last 12 months.
   3. A Papanicolaou ("Pap") smear will be required on subjects with an intact uterus and cervix if not performed within the last 6 months.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco-containing products within 1 year of start of study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial dose of study medication.
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
   3. Use hormonal replacement therapy within 3 months prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant chronic disease such as (but not limited to): 1. Thrombotic disorders. 2. Coronary artery or cerebrovascular disease. 3. Liver, kidney or gallbladder dysfunction/disorder(s). 4. Diabetes or any other endocrinological disease. 5. Estrogen-dependent neoplasia. 6. Postmenopausal uterine bleeding. 7. Endometrial hyperplasia.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, Hepatitis B, or Hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to letrozole, any of the inactive ingredients.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-11; Primary Completion 2005-12 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The 90% confidence interval for the LSMeans ratio of CPEAK, AUCL, and AUCI for the test and reference product should be between 80.00% and 125.00% for the natural log-transformed data. | Blood collections through 216 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Galitz, M.D., Principal Investigator — SFBC International
Locations (1):
- SFBC International, Miami, Florida, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html